CLINICAL TRIAL: NCT03835208
Title: The Effect of High-morning-carbohydrate Intake Versus Low-morning-carbohydrate Intake on Glycemic Variability Measured by Continuous Glucose Monitoring in GDM Patients - a Randomized Crossover Study
Brief Title: Effect of Carbohydrate Distribution on Blood Glucose in Women With Gestational Diabetes Mellitus (GDM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HMKvLMK
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-07

CONDITIONS: Diabetes, Gestational
Keywords: gestational diabetes; carbohydrate distribution; high/low carbohydrate; glycemic variability; MAGE; continuous glucose monitoring; Pregnancy in Diabetics
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy in Diabetics

STUDY DESIGN:
Intervention Model Description: Each patient will follow the HMK and LMK diet in a period of 2x3 days in randomized order with a four day washout between. The order of the two diets will be assigned randomly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-morning-carbohydrate (Experimental): Low morning intake and high evening intake of carbohydrates. This means a distribution of carbohydrate as follows:
  10% morning, 40% lunch, 50% dinner. The overall recommendations for macro- and micronutrient intake for GDM patients will be met.
  Interventions: Behavioral: High/low carbohydrate distribution
- High-morning-carbohydrate (Experimental): High morning intake and low evening intake of carbohydrates.
  This means a distribution of carbohydrate as follows:
  50% morning, 40% lunch, 10% dinner. The overall recommendations for macro- and micronutrient intake for GDM patients will be met.
  Interventions: Behavioral: High/low carbohydrate distribution

INTERVENTIONS:
Behavioral: High/low carbohydrate distribution — A total of 2x3 days, were the patient follow a detailed diet plan. For 3 days they follow a diet plan where the majority of the carbohydrates are located on either the first part of the day(HMK) or the last part of the day(LMK). 4 days of washout are placed between the two interventions. They will not receive food but will be guided by a trained dietitian and the use of a meal plan.
  Other Names: High-energy breakfasting compared with high-energy dinner

SUMMARY:
This study aims to investigate whether high-morning carbohydrate intake (HMK) compared with low-morning carbohydrate intake (LMK) affects glycemic variability in GDM patients based on Continuous glucose monitoring (CGM).

High carbohydrate morning intake is expected to reduce hyperglycemic episodes and stabilize blood glucose compared with low morning carbohydrate intake.

DETAILED DESCRIPTION:
Background:

Women with GDM have an increased risk of macrosomia, cesarean section, birth defects and long term complications such as an increased risk, in both mother and child, to develop type 2 diabetes.

According to Invitro and invivo studies of type 1 and 2 diabetes, great variations in blood glucose levels caused more complications than constantly elevated glucose levels. This study, therefore, intends to use Continuous glucose monitoring (CGM) for day-to-day monitoring of glycemic variability, including frequency, duration, and magnitude of hyperglycaemic fluctuations.

Carbohydrate is the macronutrient that has the greatest impact on postprandial blood glucose response. Despite this, there is a current lack of evidence of how the carbohydrate intake should be distributed throughout a day.

This study aims to investigate whether high-morning carbohydrate intake (HMK) compared to low-morning carbohydrate intake (LMK) affects glycemic variability in GDM patients.

Design:

Randomized crossover intervention study comparing two intervention diets; high-morning carbohydrate intake (HMK) versus low-morning carbohydrate intake (LMK) each of 3 days duration with four-day washout.

Diet intervention: Both intervention diets have the same calorie content and contain the same amounts of protein, carbohydrate and fat for the individual patient, but the distribution of carbohydrate and energy differs throughout the day.

Dietary intake will be estimated through 24-hour recall interview by trained dietitians. Estimation of actual intake is validated by photos of every main meal.

All data will be collected and stored in RedCap to secure data checks.

Statistics Analysis and sample size:

Power calculation on primary outcome MAGE- estimates 15 patients for inclusion with a power of 80%, SD 0,6mmol/l, a significance level of 0,05 and a MIREDIF of 0,5 mmol/l. 15 persons include an expected dropout rate at 20%.

Non-parametric tests will be used for the secondary and primary outcome.

Perspective:

A future perspective of this study is to improve the current treatment in regards to nutritional recommendations. Thus, the study could potentially contribute with the knowledge that would clarify the carbohydrate recommendations and improve the glycemic control of patients with GDM and therefore be beneficial to patients' future treatment and prevent complications and development of type 2 diabetes in the child.

ELIGIBILITY:
Inclusion Criteria:

* Gestational diabetes mellitus diagnosed according to current WHO criteria for a 2-hour oral glucose tolerance test (OGTT) > 8.5 mmol/l
* Non-insulin depending
* Adult 18+ years
* Gestational age weeks 30-36 at start of inclusion

Exclusion Criteria:

* Diagnosed with celiac disease
* Received bariatric surgery
* Diagnosed eating disorder
* Insulin-dependent diabetes at trial start
* Known with type 2 diabetes before pregnancy
* Children under 18 years
* Starting up in insulin during the intervention period
* Diagnosed with lactose intolerance
* Goes into labor before the intervention is completed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 15 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
mean amplitude of glucose excursions (MAGE) | 6 days
  An index for glycemic variability assessment MAGE is the average variation in amplitude and is calculated as the mean of absolute value differences between adjacent glucose peaks and valleys, where the differences exceed 1 Standard Deviation (SD) from the mean.

SECONDARY OUTCOMES:
Coefficient of variation | 6 days
  Coefficient of variation
MBG | 6 days
  The average blood glucose, calculated for each two intervention periods using CGM data.
Glucagon-like-peptide 1 (GLP1) | 1 hour *2
  glucagon-like-peptide 1, difference in 1 hour postprandial response
Gastric inhibitory polypeptide (GIP) | 1 hour*2
  Gastric inhibitory polypeptide difference in 1 hour postprandial response
C-peptide | 11 days
  Changes in C-peptide according to carbohydrate distribution

OTHER OUTCOMES:
3-hydroxy-butyrate | 11 days
  To assess ketonemia

CONTACTS AND LOCATIONS:
Overall Officials: Per G Ovesen, Dr.Med, Study Director — Women's diseases and births
Locations (2):
- Denmark (2):
  - University hospital Aarhus, Skejby, Aarhus N
  - University of Aarhus, Skejby, Aarhus N

IPD SHARING:
Plan to Share IPD: No